CLINICAL TRIAL: NCT00816036
Title: Improving the Delivery of Smoking Cessation Guidelines in Hospitalized Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Jewish Hospital Quitline (Unknown); Iowa State University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-113; NCT00962858 (obsolete NCT alias)
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-04

CONDITIONS: Cigarette Smoking
Keywords: Smoking Cessation; Practice Guidelines; Inpatient; Effectiveness Trial; Veterans Administration; Relapse prevention
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (No Intervention): Baseline Period
- Arm 2 (Experimental): Intervention Period
  Interventions: Behavioral: Smoking Cessation Guideline Implementation

INTERVENTIONS:
Behavioral: Smoking Cessation Guideline Implementation — 1. Enhanced academic detailing of staff nurses (face-to-face training, feedback on group performance, and periodic check-ins with both nurse managers and peer leaders); 2. Adaptation of the computerized information system (modified nursing admission database that includes pertinent questions about smoking, computerized "quick orders" for smoking cessation medications), 3) Patient self-management support (self-help materials, fax referral of motivated patients to state quit line), and 4) nursing peer leaders on each study unit.
  Arms: Arm 2

SUMMARY:
The primary objective of this study is to determine whether a nurse-initiated intervention, which couples brief inpatient counseling and proactive telephone counseling by a centralized tobacco quitline, improves 6-month cessation rates in hospitalized VA smokers. If proven effective, the proposed intervention will provide a practical strategy to enhance the adoption and implementation of recommended smoking cessation procedures in VA hospitals, and will demonstrate the utility of quitlines in preventing relapse in hospitalized smokers once they leave the hospital.

DETAILED DESCRIPTION:
Although the majority of hospitalized VA smokers receive some form of cessation counseling during hospitalization, few receive outpatient cessation counseling and/or pharmacotherapy following discharge, which are key factors associated with long-term cessation. The primary objective of this research study is to determine whether a nurse-initiated intervention, which couples brief inpatient counseling and proactive telephone counseling by a centralized tobacco quitline, improves 6-month cessation rates in hospitalized VA smokers. Co-primary aims are to determine whether the intervention improves the prescription of recommended pharmacotherapy for smoking cessation and the referral of patients for telephone counseling (or other outpatient cessation counseling). We will perform a quasi-experimental before-after trial in hospitalized patients, aged 18 or older, who smoke at least one cigarette per day on average. After a 6-month baseline period, we will implement the intervention and enroll a separate cohort of patients over the subsequent 6 months. The intervention will include: 1) nurse training in delivery of bedside cessation counseling, 2) use of CPRS-based practice tools (to streamline nursing assessment and documentation, to facilitate prescription of pharmacotherapy), 3) computerized referral of motivated inpatients for proactive telephone counseling, and 4) use of nursing peer leaders to provide coaching and performance feedback to ward nurses. Enrolled patients will be contacted by telephone at 3 and 6 months to assess 7-day point prevalence abstinence and prolonged abstinence (with biochemical confirmation of self-reported quitters at 6 months). We will identify barriers and facilitators to implementation by using clinician focus groups, and will assess attitudes of staff nurses toward cessation counseling by questionnaire. We will also conduct semi-structured interviews in a subsample of patients and nurses to assess perceptions of the intervention, and will use content analysis to interpret the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients: The study sample will include general medical inpatients, aged 18 or older, who smoke at least one cigarette per day on average, regardless of their willingness to quit smoking. To increase applicability of study results, the goal is to enroll patients with characteristics that reflect the full range and distribution of patients observed in clinical practice. Current smokers transferred from intensive care units (or other monitored beds) to a general medical ward will be eligible.
* Nurses: The study sample will include staff nurses who are assigned to a general medicine inpatient unit at one of the participating sites.

Exclusion Criteria:

* Hospitalization for less than 18 hours (e.g., patients admitted for overnight observation);
* Acute medical decomposition (e.g., acute respiratory failure requiring intubation, cardiac arrest, septic shock);
* Altered mental status;
* Unstable psychiatric disorder (e.g., acute psychosis);
* Dementia;
* Communication barrier (unable to speak English, hard of hearing, aphasic);
* Pregnancy;
* Terminal illness (<12 month life expectancy);
* No access to a phone or the absence of a permanent address;
* Admitted for treatment of substance abuse.

No patient will be included unless they are able to provide informed consent and agree to be contacted by telephone during follow-up (to assess smoking status).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Katz, MD MSc, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (4):
- United States (4):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Medical Center, Omaha, Omaha, Nebraska

REFERENCES:
- [Result] Katz DA, Holman J, Johnson S, Hillis SL, Ono S, Stewart K, Paez M, Fu S, Grant K, Buchanan L, Prochazka A, Battaglia C, Titler M, Vander Weg MW. Implementing smoking cessation guidelines for hospitalized veterans: effects on nurse attitudes and performance. J Gen Intern Med. 2013 Nov;28(11):1420-9. doi: 10.1007/s11606-013-2464-7. Epub 2013 May 7. PMID 23649783
- [Result] Kamath AS, Vaughan Sarrazin M, Vander Weg MW, Cai X, Cullen J, Katz DA. Hospital costs associated with smoking in veterans undergoing general surgery. J Am Coll Surg. 2012 Jun;214(6):901-8.e1. doi: 10.1016/j.jamcollsurg.2012.01.056. Epub 2012 Apr 11. PMID 22502993
- [Result] Katz D, Vander Weg M, Fu S, Prochazka A, Grant K, Buchanan L, Tinkelman D, Reisinger HS, Brooks J, Hillis SL, Joseph A, Titler M. A before-after implementation trial of smoking cessation guidelines in hospitalized veterans. Implement Sci. 2009 Sep 10;4:58. doi: 10.1186/1748-5908-4-58. PMID 19744339

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-intervention Period: Pre-intervention Period
- Intervention Period: Intervention Period
  Smoking Cessation Guideline Implementation: 1. Tutorial on brief cessation counseling for nurses and physicians; 2. use of an algorithm that includes recommended tobacco counseling items; 3. fax referral of motivated smokers to Quitline Iowa for proactive telephone counseling plus free nicotine replacement therapy; 4. group and individual feedback for staff
Period: Overall Study
Arm/Group | Pre-intervention Period | Intervention Period
Started | 503 | 395
Completed | 327 | 287
Not Completed | 176 | 108
Not completed — Death | 47 | 28
Not completed — Lost to Follow-up | 75 | 57
Not completed — Withdrawal by Subject | 54 | 23

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Pre-intervention Period
- Arm 2: Intervention Period
  Smoking Cessation Guideline Implementation: 1. Tutorial on brief cessation counseling for nurses and physicians; 2. use of an algorithm that includes recommended tobacco counseling items; 3. fax referral of motivated smokers to Quitline Iowa for proactive telephone counseling plus free nicotine replacement therapy; 4. group and individual feedback for staff
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 503 | 395 | 898
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.7) | 58.8 (10.2) | 59.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 36
  Male | 480 | 382 | 862
Region of Enrollment [Number; unit: participants]
  United States | 503 | 395 | 898

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point-prevalence Smoking Abstinence (6-month)
Description: This is the number of patients who reported not have smoked cigarettes over the 7 days prior to the 6-month follow-up interview.
Time Frame: 6 months post enrollment
Population: This is the total number of subjects who completed 6 month follow-up (complete case analysis).
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 498 | 394
participants | 69 | 53

2. Secondary Outcome: Referrals to Quitline
Time Frame: Assessed within 72 hours of hospital discharge
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 498 | 394
participants | 0 | 36

3. Secondary Outcome: Prescription of Recommended Pharmacotherapy for Smoking Cessation
Time Frame: Assessed within 72 hours of hospital discharge
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 498 | 394
participants | 176 | 149

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/503 | 0/395
Other Adverse Events (participants affected / at risk) | 0/503 | 0/395

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes